CLINICAL TRIAL: NCT03350867
Title: Effects of Using Customized Insoles With Anterior or Posterior Plantar Support in Cross-pelvis Syndrome and Perception of Body Alignment in Young Adults: a Randomized Clinical Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidade Federal de Pernambuco (Other)
Responsible Party: Principal Investigator, Eduardo Augusto dos Santos Pimentel, Eduardo Augusto Dos Santos Pimentel, Universidade Federal de Pernambuco
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Insole and cross-pelvis synd.
Record Dates: First submitted 2017-11-18; First posted 2017-11-22 (Actual); Last update posted 2017-11-22 (Actual); Status verified 2017-11

CONDITIONS: Crossed Pelvis Syndrome
Keywords: Posture; Orthosis; Foot; Biomechanical Phenomena

STUDY DESIGN:
Intervention Model Description: Two groups: a Personalized Insole Group and a Placebo Group.
Who Masked: Participant, Outcomes Assessor
Masking Description: Double (Participant, Outcomes Assessor) The one who assess the patients in the beginning and in the final moment (investigator) not know what group the patient is. The participants don't know if they are using a placebo or personalized insole.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Personalized Insole Group (Experimental): The participants will use insole with personalized support directed to your biomechanics necessities.
  Interventions: Other: Personalized Insole Group
- Placebo Group (Placebo Comparator): The participants will use plane insoles.
  Interventions: Other: Placebo Group

INTERVENTIONS:
Other: Personalized Insole Group — Personalized Insole Group
  Arms: Personalized Insole Group
Other: Placebo Group — Placebo Group
  Arms: Placebo Group

SUMMARY:
INTRODUCTION: Custom insoles with anterior or posterior support are described in the literature mainly for the treatment of foot and knee dysfunctions and this therapeutic effect extends to the promotion of biomechanical alignment between pelvis and trunk, by an ascending propceptive response. In this perspective, it can be hypothesized that the use of these insoles may favor individuals with anterior and posterior cross pelvis syndrome, who have biomechanical imbalance in the pelvis segment. To date, there is no literature data on the effect of continuous, noninvasive and inexpensive therapy on this individual profile.

OBJECTIVE: To evaluate the effects of using customized insoles with anterior or posterior plantar support in cross pelvis syndrome and in perception of body alignment in young adults.

METHODS: This is a blinded randomized controlled trial in individuals of both sexes aged 18-25 years and functionally diagnosed with posterior or anterior pelvic syndrome. Excluding thoracic deformities, lower limb differences, diabetic neuropathy, previous reports of some specific surgeries and treatment of ongoing physiotherapy. A pilot study will be carried out with 20 individuals divided into two groups for sample calculation (Personalized Insole Group and Placebo Group). After the pilot study, an initial screening will be carried out to verify the eligibility criteria. For the eligible, the pre-intervention evaluation will be carried out, which will be contemplated by personal data; scale of presence and intensity of pain; foot health status; foot posture index; by ely and thomas hamstring tests associated with an inclinometer and by photogrammetry. Individuals will be randomized into blocks of 10 individuals. A day will be marked to make the insole, in which the researcher will make the adaptations based on the biomechanical evaluation of the volunteer. To the invidious with the posterior cross pelvis syndrome an anterior support will be made in the insole and for those with anterior cross pelvis syndrome a posterior support will be made in the insole. For the placebo group, the insole will be made of the same material as that of the custom insoles, although, without support.

ELIGIBILITY:
Inclusion Criteria:

* Crossed pelvis syndrome (anterior or posterior)
* Difference in length leg ≤ 1cm
* Don't show: scoliotic or kyphotic deformity; chirurgie or fracture in spine in last 12 months; thoracic chirurgie; diabetic neuropathy; cesarean surgery; mixed crossed pelvis syndrome
* Not participating in any physical activity or physiotherapy

Exclusion Criteria:

* Join in other physical activity during the study
* Refuse to wear the insoles

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Estimated)
Dates: Start 2017-08-09 (Actual); Primary Completion 2017-12-20 (Estimated); Study Completion 2017-12-20 (Estimated)

PRIMARY OUTCOMES:
Posture | 45 days
  Photogrammetry in Corel Draw

SECONDARY OUTCOMES:
Pain | 45 days
  Visual analog scale.
Moviment amplitude (hip joint, knee) | 45 days
  Goniometry
Lombar colune mobility | 45 days
  Schober test
Abdominal circunference | 45 days
  Roma test
Sacroiliac mobility | 45 days
  Standing flexion test and Gillet test

CONTACTS AND LOCATIONS:
Locations (1):
- Laboratory of learning and motor control; Federal University of Pernambuco (UFPE), Recife, Pernambuco, Brazil